CLINICAL TRIAL: NCT02626286
Title: Prevention of HIV Infection in Men Who Have Sex With Men in Sub-Saharan Africa: Feasibility and Interest of a Quarterly Preventive Global Care (CohMSM)
Brief Title: Feasibility and Interest of a HIV Quarterly Preventive Global Care in Men Who Have Sex With Men in Sub-Saharan Africa
Acronym: CohMSM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: ANRS, Emerging Infectious Diseases (Other Government)
Collaborators: Expertise France (Other); Université Montpellier (Other); IRD Unité SESSTIM (IRD, Inserm, Université Aix-Marseille) (Unknown); Coalition Internationale Sida (Other); ARCAD-SIDA MALI (Other); Espace Confiance, Côte d'Ivoire (Other); Programme PAC-CI, Abidjan, Côte d'Ivoire (Unknown); Association African Solidarité (Other); Centre de Recherche Internationale pour la Santé, Ouagadougou, Burkina Faso (Unknown); Espoir Vie-Togo - ONG (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: ANRS 12324 CohMSM
Record Dates: First submitted 2015-11-20; First posted 2015-12-10 (Estimated); Last update posted 2021-04-22 (Actual); Status verified 2021-04

CONDITIONS: HIV Infection
Keywords: HIV; Men who have sex with men
MeSH Terms: conditions — HIV Infections; Homosexuality

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- HIV quarterly global care (Other): HIV quarterly global care including i) data collection on health status, symptoms of sexually transmitted infections (STI) and sexual behavior, ii) a clinical examination, iii) STI diagnosis and treatment, iv) prevention counselling adapted for MSM, v) the provision of condoms and lubricants, and vi) HIV screening test at each quarterly visit for HIV-negative MSM or immediate support of HIV infection including antiretroviral therapy for HIV-positive MSM.
  Interventions: Other: HIV quarterly global care

INTERVENTIONS:
Other: HIV quarterly global care

SUMMARY:
The objective of the study is to evaluate the feasibility and interest of a HIV quarterly preventive global care for men who have sex with men (MSM) in sub-Saharan Africa to help reducing HIV incidence in this key population, their female partners, and the general population. This interventional, open label, multicenter, multidisciplinary cohort study will be conducted in Burkina Faso, Ivory Coast, Mali and Togo.

All participants will receive a HIV quarterly preventive global care including:

i) data collection on health status, symptoms of sexually transmitted infections (STI) and sexual behavior, ii) a clinical examination, iii) STI diagnosis and treatment, iv) counselling adapted for MSM, and v) the provision of condoms and lubricants.

DETAILED DESCRIPTION:
The objective of the study is to evaluate the feasibility and interest of a HIV quarterly preventive global care for men who have sex with men (MSM) in sub-Saharan Africa to help reducing HIV incidence in this key population, their female partners, and the general population.

Regarding HIV-negative MSM, the specific objectives are to assess:

1. the acceptability of the preventive global care including quarterly monitoring and HIV screening as well as the associated medical, behavioral and social factors, and
2. changes in sexual behavior among MSM during the project as well as the associated medical, behavioral and social factors.

Regarding HIV-positive MSM, the specific objectives are to assess:

1. the acceptability of the preventive global care including antiretroviral therapy initiation whatever the CD4 T cell count and the clinical stage, as well as the associated medical, behavioral and social factors,
2. adherence and response to antiretroviral therapy as well as the associated medical, behavioral and social factors,
3. changes in sexual behavior among MSM during the project as well as the associated medical, behavioral and social factors,
4. risk of HIV transmission as well as the associated medical, behavioral and social factors, and
5. describe the virologic characteristics (subtypes / circulating recombinant forms, co-infection with multiple variants and transmitted and acquired resistance profiles).

Regarding healthcare professionals, the specific objective is to evaluate the perception of the preventive global care.

This interventional, open label, multicenter, multidisciplinary cohort study will be conducted in Burkina Faso, Ivory Coast, Mali and Togo.

All participants will receive a HIV quarterly preventive global care including:

i) data collection on health status, symptoms of sexually transmitted infections (STI) and sexual behavior, ii) a clinical examination, iii) STI diagnosis and treatment, iv) counselling adapted for MSM, and v) the provision of condoms and lubricants.

In addition, vaccination against hepatitis B virus and annual tests for syphilis will be offered. HIV-negative MSM will also be offered an HIV screening test at each quarterly visit. HIV-positive MSM will be offered immediate support of HIV infection including antiretroviral therapy. A total of 700 MSM over 18 years (500 HIV-negative and 200 HIV-positive) reporting at least one anal sex (passive or active) with another man within the last three months will be recruited and followed for 24 to 36 months. MSM lost to follow-up, transferred, died or having seroconverted for HIV during follow-up will be replaced in their respective group (seronegative or seropositive) by other MSM. The study will last 3 years.

ELIGIBILITY:
Inclusion Criteria:

* Man over 18 years
* Reporting at least one anal sex (passive or active) with another man within the last three months
* Able to reach the local site of the study
* Agreeing to participate in the study and signing the informed consent form

Exclusion Criteria:

* History of antiretroviral therapy (except for pre- or post-exposure prophylaxis)
* Participation in another biomedical or behavioral research on HIV or sexually transmitted infections
* Impairment of the person making his participation in the study, or information understanding, difficult or impossible
* Predictable protocol violation (geographical distance or other reasons)

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 885 (Actual)
Dates: Start 2015-06 (Actual); Primary Completion 2021-01-05 (Actual); Study Completion 2021-01-05 (Actual)

PRIMARY OUTCOMES:
Number of people followed after 3 years compared to the number of persons included (retention in the program) | 3 years
Percentage of performed visits/scheduled visits | 3 years
Percentage of performed tests/scheduled tests | 3 years
Incidence of sexually transmitted infections | 3 years
Number of unprotected anal sex | 3 years
Antiretroviral therapy initiation probability in HIV-positive MSM | 3 years
Antiretroviral therapy maintenance probability in HIV-positive MSM | 3 years
Percentage of antiretroviral therapy observance in HIV-positive MSM | 3 years
Percentage of HIV-positive MSM with viral load>1000 copies/mL | 3 years
Percentage of HIV-positive MSM with CD4≤reference (or CD4<100/mm3) | 3 years
Percentage of HIV-positive MSM with new or recurrent AIDS-defining events (clinical stage 4) | 3 years
Percentage of HIV-positive MSM died under antiretroviral therapy | 3 years
Percentage of HIV-positive MSM with detectable viral load and inconsistent condom use with a partner seronegative or with unknown HIV status | 3 years
Number of HIV subtypes / circulating recombinant forms | 3 years
Number of co-infections with several viral variants | 3 years
Number of transmitted and acquired resistance mutations | 3 years
Number of male sex partners | 3 years

CONTACTS AND LOCATIONS:
Locations (4):
- Centre Oasis, Association African Solidarité (AAS), Ouagadougou, Burkina Faso
- Clinique de Confiance, Espace Confiance, Abidjan, Côte d’Ivoire
- Clinique des Halles, ARCAD-SIDA, Bamako, Mali
- Espoir vie Togo, Lomé, Togo

REFERENCES:
- [Derived] Dah TTE, Yaya I, Mensah E, Coulibaly A, Kouame JM, Traore I, Mora M, Palvadeau P, Anoma C, Keita BD, Spire B, Laurent C; CohMSM Study Group. Rapid antiretroviral therapy initiation and its effect on treatment response in MSM in West Africa. AIDS. 2021 Nov 1;35(13):2201-2210. doi: 10.1097/QAD.0000000000003046. PMID 34352834
- [Derived] Dah TTE, Yaya I, Sagaon-Teyssier L, Coulibaly A, Kouame MJ, Agboyibor MK, Maiga K, Traore I, Mora M, Palvadeau P, Rojas-Castro D, Diallo F, Mensah E, Anoma C, Keita BD, Spire B, Laurent C; CohMSM Study Group. Adherence to quarterly HIV prevention services and its impact on HIV incidence in men who have sex with men in West Africa (CohMSM ANRS 12324 - Expertise France). BMC Public Health. 2021 May 22;21(1):972. doi: 10.1186/s12889-021-10994-4. PMID 34022820
- [Derived] Yaya I, Diallo F, Kouame MJ, Agboyibor MK, Traore I, Coulibaly A, Maiga K, Mora M, Palvadeau P, Dah ETT, Mensah E, Anoma C, Dembele Keita B, Spire B, Laurent C; CohMSM Study Group. Decrease in incidence of sexually transmitted infections symptoms in men who have sex with men enrolled in a quarterly HIV prevention and care programme in West Africa (CohMSM ANRS 12324-Expertise France). Sex Transm Infect. 2022 Mar;98(2):85-94. doi: 10.1136/sextrans-2020-054755. Epub 2021 Mar 22. PMID 33753460